CLINICAL TRIAL: NCT03438383
Title: The Effect of Bi-PAP at Individualized Pressures on the Postoperative Pulmonary Recovery of Morbidly Obese Patients (MOP) Undergoing Open Bariatric Surgery (OBS) and Possible Placebo Device-related Effects (Sham-Bi-PAP)
Brief Title: Bi-PAP vs Sham Bi-PAP on Pulmonary Function in Morbidly Obese Patients After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Collaborators: Elpis General Hospital (Unknown); Sotiria General Hospital (Other); Evgenidion Hospital (Unknown)
Responsible Party: Principal Investigator, Alexandropoulou N. Aikaterini, Consultant, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 142/23-05-2011
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Atelectasis; Pulmonary Infection; Chronic Obstructive Pulmonary Disease (COPD); Pulmonary Disease; Hypoxemic Respiratory Failure; Hypoxemia; Morbid Obesity
Keywords: Bi-PAP; BiPAP; morbid obesity; anesthesia; bariatric surgery; sham Bi-PAP; sham BiPAP; postoperative complications
MeSH Terms: conditions — Pulmonary Atelectasis; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Insufficiency; Hypoxia; Obesity, Morbid; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Patients were assigned into the following two study groups postoperatively:
  1. Sham Bi-PAP (control group) group in which sham Bi-PAP was applied through nasal mask for 3 days postoperatively.
  2. Bi-PAP group in which Bi-PAP through nasal mask, at individualized IPAP/EPAP pressures, was applied for 3 days postoperatively.
  1 patient was initially enrolled in the protocol but was excluded from the participant flow design because of recent onset of cardiovascular disease (CAD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham Bi-PAP (Sham Comparator): Sham Bi-PAP was applied through nasal mask for 3 days postoperatively. Sham Bi-PAP was created by introducing a "hole" at the connection of the mask with the spiral tube of Bi-PAP. With this modality, also used on previous studies, the applied pressure by sham Bi-PAP was constant and equal to 2 centimeter of water (cm H2O).
  Interventions: Device: Sham Bi-PAP
- Bi-PAP (Active Comparator): Bi-PAP through nasal mask, at individualized IPAP/EPAP pressures, was applied for 3 days postoperatively. IPAP and EPAP in the Bi-PAP system were individualized for each patient in accordance with accepted values of SpO2, PaCO2, and patient synchronization and tolerability with the device.Individualized setting of pressures in patient group was applied gradually starting with 12/4 cm H2O (IPAP/EPAP) and up to 18/10 (IPAP/EPAP) with consecutive increases of 2 cm H2O.
  Interventions: Device: Bi-PAP

INTERVENTIONS:
Device: Bi-PAP — The Bi-PAP system combines inspiratory support-IPAP (inspiratory positive airway pressure) with expiratory support-EPAP (expiratory positive airway pressure) and has been used, with good results, in a number of different clinical conditions such as COPD, respiratory failure due to neuromuscular disease, cardiogenic pulmonary edema and immediately post-operatively with pro-phylactic purpose.
  Arms: Bi-PAP
Device: Sham Bi-PAP — Sham Bi-PAP was created by introducing a "hole" at the connection of the mask with the spiral tube of the conventional Bi-PAP system. By doing so, the applied pressure by sham Bi-PAP was constant and equal to 2 cm H2O.
  Arms: Sham Bi-PAP

SUMMARY:
The effect of biphasic positive airway pressure (Bi-PAP) at individualized pressures on the postoperative pulmonary recovery of morbidly obese patients (MOP) undergoing open bariatric surgery (OBS) and possible placebo device-related effects (sham-Bi-PAP) were investigated.

DETAILED DESCRIPTION:
In the present study the effect of Bi-PAP on the postoperative respiratory function and related complications of MOP undergoing OBS through a randomized sham-controlled design was investigated. Bi-PAP was applied at individualized pressures in order to optimize respiratory support and sham Bi-PAP was also used in order to neutralize possible placebo device related effect and researcher related bias.

The investigators hypothesized that the use of Bi-PAP at individualized pressures in MOP undergoing OBS, ameliorates postoperative respiratory function as well as diminishes related pulmonary complications, postoperative pain and duration of hospitalization. Primary endpoints were the difference in pre- and postoperative measurements of certain pulmonary function parameters (forced expiratory volume at one second (FEV1), forced vital capacity (FVC), peak expiratory flow rate (PEFR) and oxygen saturation by pulse oximetry (SpO2) and the incidence of certain pulmonary complications postoperatively (hypoxemia, atelectasis, lower respiratory tract infections). Secondary endpoints were postoperative pain and days of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* All patients have been Morbidly Obese (BMI> 40kg/m2) for at least 10 years
* All patients had unsuccessfully tried to lose weight by other non-invasive means.
* All patients enrolled were continuous positive airway pressure (CPAP) and Bi-PAP naïve and had no knowledge about the Bi-PAP apparatus prior to enrollment
* All patients underwent OBS (gastroplasty by Mason or gastric bypass) by the same operating team
* All patients were treated with the same standard anesthetic protocol

Exclusion Criteria:

* Cardiovascular and pulmonary disease not related to obesity status
* Chronic renal disease
* Patients who were initially enrolled but did not use the allocated device (Bi-PAP or Sham Bi-PAP) for at least 12 h daily were also excluded at a later point.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2012-05-22 (Actual); Study Completion 2012-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Louis, MD, PhD, Study Director — Dpt of ObGyn, Konstantopoulio-Patision Hospital, Greece; Konstantinos Roditis, MD, MSc, Study Chair — Dpt of Vascular Surgery, Korgialenio-Benakio HRC Hospital, Greece; Aikaterini N. Alexandropoulou, MD, PhD, Principal Investigator — Anaesthesiology Dpt, Evangelismos Hospital, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parameswaran K, Todd DC, Soth M. Altered respiratory physiology in obesity. Can Respir J. 2006 May-Jun;13(4):203-10. doi: 10.1155/2006/834786. PMID 16779465
- [Background] Salome CM, King GG, Berend N. Physiology of obesity and effects on lung function. J Appl Physiol (1985). 2010 Jan;108(1):206-11. doi: 10.1152/japplphysiol.00694.2009. Epub 2009 Oct 29. PMID 19875713
- [Background] Gifford AH, Leiter JC, Manning HL. Respiratory function in an obese patient with sleep-disordered breathing. Chest. 2010 Sep;138(3):704-15. doi: 10.1378/chest.09-3030. No abstract available. PMID 20822992
- [Background] Littleton SW. Impact of obesity on respiratory function. Respirology. 2012 Jan;17(1):43-9. doi: 10.1111/j.1440-1843.2011.02096.x. PMID 22040049
- [Background] Hans GA, Lauwick S, Kaba A, Brichant JF, Joris JL. Postoperative respiratory problems in morbidly obese patients. Acta Anaesthesiol Belg. 2009;60(3):169-75. PMID 19961114
- [Background] Lawrence VA, Dhanda R, Hilsenbeck SG, Page CP. Risk of pulmonary complications after elective abdominal surgery. Chest. 1996 Sep;110(3):744-50. doi: 10.1378/chest.110.3.744. PMID 8797421
- [Background] Simonneau G, Vivien A, Sartene R, Kunstlinger F, Samii K, Noviant Y, Duroux P. Diaphragm dysfunction induced by upper abdominal surgery. Role of postoperative pain. Am Rev Respir Dis. 1983 Nov;128(5):899-903. doi: 10.1164/arrd.1983.128.5.899. PMID 6638679
- [Background] Vassilakopoulos T, Mastora Z, Katsaounou P, Doukas G, Klimopoulos S, Roussos C, Zakynthinos S. Contribution of pain to inspiratory muscle dysfunction after upper abdominal surgery: A randomized controlled trial. Am J Respir Crit Care Med. 2000 Apr;161(4 Pt 1):1372-5. doi: 10.1164/ajrccm.161.4.9907082. PMID 10764336
- [Background] Pelosi P, Gregoretti C. Perioperative management of obese patients. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):211-25. doi: 10.1016/j.bpa.2010.02.001. PMID 20608558
- [Background] Loadsman JA, Hillman DR. Anaesthesia and sleep apnoea. Br J Anaesth. 2001 Feb;86(2):254-66. doi: 10.1093/bja/86.2.254. PMID 11573670
- [Background] Cullen A, Ferguson A. Perioperative management of the severely obese patient: a selective pathophysiological review. Can J Anaesth. 2012 Oct;59(10):974-96. doi: 10.1007/s12630-012-9760-2. Epub 2012 Jul 26. PMID 22833138
- [Background] Casati A, Putzu M. Anesthesia in the obese patient: pharmacokinetic considerations. J Clin Anesth. 2005 Mar;17(2):134-45. doi: 10.1016/j.jclinane.2004.01.009. PMID 15809132
- [Background] Kyzer S, Ramadan E, Gersch M, Chaimoff C. Patient-Controlled Analgesia Following Vertical Gastroplasty: a Comparison with Intramuscular Narcotics. Obes Surg. 1995 Feb;5(1):18-21. doi: 10.1381/096089295765558097. PMID 10733789
- [Background] Charghi R, Backman S, Christou N, Rouah F, Schricker T. Patient controlled i.v. analgesia is an acceptable pain management strategy in morbidly obese patients undergoing gastric bypass surgery. A retrospective comparison with epidural analgesia. Can J Anaesth. 2003 Aug-Sep;50(7):672-8. doi: 10.1007/BF03018709. PMID 12944441
- [Background] Nguyen NT, Lee SL, Goldman C, Fleming N, Arango A, McFall R, Wolfe BM. Comparison of pulmonary function and postoperative pain after laparoscopic versus open gastric bypass: a randomized trial. J Am Coll Surg. 2001 Apr;192(4):469-76; discussion 476-7. doi: 10.1016/s1072-7515(01)00822-5. PMID 11294404
- [Background] Thomas JA, McIntosh JM. Are incentive spirometry, intermittent positive pressure breathing, and deep breathing exercises effective in the prevention of postoperative pulmonary complications after upper abdominal surgery? A systematic overview and meta-analysis. Phys Ther. 1994 Jan;74(1):3-10; discussion 10-6. doi: 10.1093/ptj/74.1.3. PMID 8265725
- [Background] Ambrosino N, Gabbrielli L. Physiotherapy in the perioperative period. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):283-9. doi: 10.1016/j.bpa.2010.02.003. PMID 20608563
- [Background] Mehta S, Hill NS. Noninvasive ventilation. Am J Respir Crit Care Med. 2001 Feb;163(2):540-77. doi: 10.1164/ajrccm.163.2.9906116. No abstract available. PMID 11179136
- [Background] Pelosi P, Jaber S. Noninvasive respiratory support in the perioperative period. Curr Opin Anaesthesiol. 2010 Apr;23(2):233-8. doi: 10.1097/ACO.0b013e328335daec. PMID 20019602
- [Background] Renston JP, DiMarco AF, Supinski GS. Respiratory muscle rest using nasal BiPAP ventilation in patients with stable severe COPD. Chest. 1994 Apr;105(4):1053-60. doi: 10.1378/chest.105.4.1053. PMID 8162724
- [Background] Radunovic A, Annane D, Rafiq MK, Mustfa N. Mechanical ventilation for amyotrophic lateral sclerosis/motor neuron disease. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD004427. doi: 10.1002/14651858.CD004427.pub3. PMID 23543531
- [Background] Nava S, Carbone G, DiBattista N, Bellone A, Baiardi P, Cosentini R, Marenco M, Giostra F, Borasi G, Groff P. Noninvasive ventilation in cardiogenic pulmonary edema: a multicenter randomized trial. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1432-7. doi: 10.1164/rccm.200211-1270OC. Epub 2003 Sep 4. PMID 12958051
- [Background] Moritz F, Brousse B, Gellee B, Chajara A, L'Her E, Hellot MF, Benichou J. Continuous positive airway pressure versus bilevel noninvasive ventilation in acute cardiogenic pulmonary edema: a randomized multicenter trial. Ann Emerg Med. 2007 Dec;50(6):666-75, 675.e1. doi: 10.1016/j.annemergmed.2007.06.488. Epub 2007 Aug 30. PMID 17764785
- [Background] Gust R, Gottschalk A, Schmidt H, Bottiger BW, Bohrer H, Martin E. Effects of continuous (CPAP) and bi-level positive airway pressure (BiPAP) on extravascular lung water after extubation of the trachea in patients following coronary artery bypass grafting. Intensive Care Med. 1996 Dec;22(12):1345-50. doi: 10.1007/BF01709549. PMID 8986484
- [Background] Aguilo R, Togores B, Pons S, Rubi M, Barbe F, Agusti AG. Noninvasive ventilatory support after lung resectional surgery. Chest. 1997 Jul;112(1):117-21. doi: 10.1378/chest.112.1.117. PMID 9228366
- [Background] Joris JL, Sottiaux TM, Chiche JD, Desaive CJ, Lamy ML. Effect of bi-level positive airway pressure (BiPAP) nasal ventilation on the postoperative pulmonary restrictive syndrome in obese patients undergoing gastroplasty. Chest. 1997 Mar;111(3):665-70. doi: 10.1378/chest.111.3.665. PMID 9118706
- [Background] Ebeo CT, Benotti PN, Byrd RP Jr, Elmaghraby Z, Lui J. The effect of bi-level positive airway pressure on postoperative pulmonary function following gastric surgery for obesity. Respir Med. 2002 Sep;96(9):672-6. doi: 10.1053/rmed.2002.1357. PMID 12243311
- [Background] Soroksky A, Stav D, Shpirer I. A pilot prospective, randomized, placebo-controlled trial of bilevel positive airway pressure in acute asthmatic attack. Chest. 2003 Apr;123(4):1018-25. doi: 10.1378/chest.123.4.1018. PMID 12684289
- [Background] Thys F, Roeseler J, Reynaert M, Liistro G, Rodenstein DO. Noninvasive ventilation for acute respiratory failure: a prospective randomised placebo-controlled trial. Eur Respir J. 2002 Sep;20(3):545-55. doi: 10.1183/09031936.02.00287402. PMID 12358327
- [Background] Crapo RO. Pulmonary-function testing. N Engl J Med. 1994 Jul 7;331(1):25-30. doi: 10.1056/NEJM199407073310107. No abstract available. PMID 8202099
- [Background] Lumb AB, Greenhill SJ, Simpson MP, Stewart J. Lung recruitment and positive airway pressure before extubation does not improve oxygenation in the post-anaesthesia care unit: a randomized clinical trial. Br J Anaesth. 2010 May;104(5):643-7. doi: 10.1093/bja/aeq080. Epub 2010 Mar 30. PMID 20354010
- [Background] Neligan PJ, Malhotra G, Fraser M, Williams N, Greenblatt EP, Cereda M, Ochroch EA. Continuous positive airway pressure via the Boussignac system immediately after extubation improves lung function in morbidly obese patients with obstructive sleep apnea undergoing laparoscopic bariatric surgery. Anesthesiology. 2009 Apr;110(4):878-84. doi: 10.1097/ALN.0b013e31819b5d8c. PMID 19293693
- [Background] Wong DT, Adly E, Ip HY, Thapar S, Maxted GR, Chung FF. A comparison between the Boussignac continuous positive airway pressure mask and the venturi mask in terms of improvement in the PaO2/F(I)O2 ratio in morbidly obese patients undergoing bariatric surgery: a randomized controlled trial. Can J Anaesth. 2011 Jun;58(6):532-9. doi: 10.1007/s12630-011-9497-3. Epub 2011 Apr 5. PMID 21465320
- [Background] Cobbold A, Lord S. Treatment and management of obesity: is surgical intervention the answer? J Perioper Pract. 2012 Apr;22(4):114-21. doi: 10.1177/175045891202200404. PMID 22567762
- [Background] Talab HF, Zabani IA, Abdelrahman HS, Bukhari WL, Mamoun I, Ashour MA, Sadeq BB, El Sayed SI. Intraoperative ventilatory strategies for prevention of pulmonary atelectasis in obese patients undergoing laparoscopic bariatric surgery. Anesth Analg. 2009 Nov;109(5):1511-6. doi: 10.1213/ANE.0b013e3181ba7945. PMID 19843790
- [Background] Eichenberger A, Proietti S, Wicky S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Morbid obesity and postoperative pulmonary atelectasis: an underestimated problem. Anesth Analg. 2002 Dec;95(6):1788-92, table of contents. doi: 10.1097/00000539-200212000-00060. PMID 12456460
- [Background] Ramirez A, Lalor PF, Szomstein S, Rosenthal RJ. Continuous positive airway pressure in immediate postoperative period after laparoscopic Roux-en-Y gastric bypass: is it safe? Surg Obes Relat Dis. 2009 Sep-Oct;5(5):544-6. doi: 10.1016/j.soard.2009.05.007. Epub 2009 Jun 23. PMID 19640798
- [Background] Vasquez TL, Hoddinott K. A potential complication of bi-level positive airway pressure after gastric bypass surgery. Obes Surg. 2004 Feb;14(2):282-4. doi: 10.1381/096089204322857717. PMID 15018761
- [Background] Huerta S, DeShields S, Shpiner R, Li Z, Liu C, Sawicki M, Arteaga J, Livingston EH. Safety and efficacy of postoperative continuous positive airway pressure to prevent pulmonary complications after Roux-en-Y gastric bypass. J Gastrointest Surg. 2002 May-Jun;6(3):354-8. doi: 10.1016/s1091-255x(01)00048-8. PMID 12022987
- [Result] Alexandropoulou AN, Louis K, Papakonstantinou A, Tzirogiannis K, Stamataki E, Roussos C, Alchanatis M, Gratziou C, Vagiakis E, Roditis K. The influence of biphasic positive airway pressure vs. sham biphasic positive airway pressure on pulmonary function in morbidly obese patients after bariatric surgery. Anaesthesiol Intensive Ther. 2019;51(2):88-95. doi: 10.5114/ait.2019.85868. PMID 31268268
- See also: Publication of Study Results — https://www.termedia.pl/Journal/-118/pdf-36902-10?filename=The%20influence%20of%20biphasic.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Τhis prospective randomized single-blinded study with a control group was conducted in a tertiary urban Greek hospital. Subjects recruitment was performed at the respective departments of obesity surgery where subjects underwent surgery, also belonging to tertiary hospitals.
Pre-assignment Details: Exclusion criteria included cardiovascular and pulmonary disease not related to obesity status, and chronic renal disease. From the 48 patients initially enrolled in the study, 1 was excluded from the participant flow because of recent onset of cardiovascular disease. 47 patients were assigned to the study groups.
Groups:
- Sham Bi-PAP: Sham Bi-PAP was applied through nasal mask for 3 days postoperatively. Sham Bi-PAP was created by introducing a "hole" at the connection of the mask with the spiral tube of Bi-PAP. With this modality, also used on previous studies, the applied pressure by sham Bi-PAP was constant and equal to 2 centimeters of water (cm H2O).
  Sham Bi-PAP: Sham Bi-PAP was created by introducing a "hole" at the connection of the mask with the spiral tube of the conventional Bi-PAP system. By doing so, the applied pressure by sham Bi-PAP was constant and equal to 2 cm H2O.
- Bi-PAP: Bi-PAP through nasal mask, at individualized IPAP/EPAP pressures, was applied for 3 days postoperatively. IPAP and EPAP in the Bi-PAP system were individualized for each patient in accordance with accepted values of oxygen saturation by pulse oximetry (SpO2), PaCO2, and patient synchronization and tolerability with the device.Individualized setting of pressures in patient group was applied gradually starting with 12/4 cm H2O (IPAP/EPAP) and up to 18/10 (IPAP/EPAP) with consecutive increases of 2 cm H2O.
  Bi-PAP: The Bi-PAP system combines inspiratory support-IPAP (inspiratory positive airway pressure) with expiratory support-EPAP (expiratory positive airway pressure) and has been used, with good results, in a number of different clinical conditions such as chronic obstructive pulmonary disease (COPD), respiratory failure due to neuromuscular disease, cardiogenic pulmonary edema and immediately post-operatively with pro-phylactic purpose.
Period: Overall Study
Arm/Group | Sham Bi-PAP | Bi-PAP
Started | 23 | 24
Completed | 14 | 21
Not Completed | 9 | 3
Not completed — Protocol Violation | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sham Bi-PAP: Sham Bi-PAP was applied through nasal mask for 3 days postoperatively. Sham Bi-PAP was created by introducing a "hole" at the connection of the mask with the spiral tube of Bi-PAP. With this modality, also used on previous studies, the applied pressure by sham Bi-PAP was constant and equal to 2 cm H2O.
  Sham Bi-PAP: Sham Bi-PAP was created by introducing a "hole" at the connection of the mask with the spiral tube of the conventional Bi-PAP system. By doing so, the applied pressure by sham Bi-PAP was constant and equal to 2 cm H2O.
- Total: Total of all reporting groups
Arm/Group | Sham Bi-PAP | Bi-PAP | Total
Number analyzed (Participants) | 14 | 21 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8) | 31 (6) | 31.8 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 21 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 21 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 14 | 21 | 35
Height [Mean (Standard Deviation); unit: Centimeters] | 171 (7) | 172 (27) | 171.6 (21.16)
Weight [Mean (Standard Deviation); unit: Kilograms] | 151 (30) | 157 (27) | 154.6 (27.96)
Body mass index-BMI [Mean (Standard Deviation); unit: Kilograms/squared meters] | 52 (6) | 53 (8) | 52.6 (7.19)
Smoking [Count of Participants; unit: Participants] — Whether the subject declared as an active smoker
  Participants | 7 | 14 | 21
Type of open bariatric surgery (OBS): gastroplasty [Count of Participants; unit: Participants] | 11 | 15 | 26
Type of OBS: open gastric bypass [Count of Participants; unit: Participants] | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume at One Second (FEV1) Difference
Description: difference in FEV1 value measured by spirometry pre- and post-operatively
Time Frame: 24 h before surgery and at 24, 48 and 72 h post-operatively
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
Litres
  24h before surgery | 3.1 (0.7) | 3.1 (0.6)
  24h post-op | 1.3 (0.5) | 1.4 (0.3)
  48h post-op | 1.3 (0.4) | 1.7 (0.4)
  72h post-op | 1.4 (0.5) | 1.9 (0.4)
Statistical Analysis 1: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h before surgery (pre-operative or baseline values); Test type: Superiority — We computed (post-hoc) the observed power of the performed tests (ANOVA for repeated measures). We confirmed that the specific sample size, as calculated using the Do-it-Yourself (DiY) sample size calculator (online at: https://blog.exmr.net/ sample-size-calculator) by considering a confidence level of 95% and a 10% margin of error, yielded adequate statistical power (> 80%) for each of the examined variables; p = 0.88, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 2: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.23, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 3: Comparison: Sham Bi-PAP vs Bi-PAP; 48 hours post-operatively; Test type: Superiority — We checked for equivalence of the pre-op (baseline) values between the two groups. We computed (post-hoc) the observed power of the performed tests (ANOVA for repeated measures). We confirmed that the specific sample size, as calculated using the Do-it-Yourself (DiY) sample size calculator (online at: https://blog.exmr.net/ sample-size-calculator) by considering a confidence level of 95% and a 10% margin of error, yielded adequate statistical power (> 80%) for each of the examined variables; p = 0.008, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 4: Comparison: Sham Bi-PAP vs Bi-PAP; 72 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.001, ANOVA — The a priori threshold for statistical significance was set at <0.05

2. Primary Outcome: Forced Vital Capacity (FVC) Difference
Description: difference in FVC value measured by spirometry pre- and post-operatively
Time Frame: 24 h before surgery and at 24, 48 and 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
Litres
  24h before surgery | 3.4 (1.0) | 3.5 (0.7)
  24h post-op | 1.3 (0.4) | 1.6 (0.4)
  48h post-op | 1.5 (0.5) | 2.0 (0.4)
  72h post-op | 1.9 (0.6) | 2.3 (0.4)
Statistical Analysis 1: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h before surgery (pre-operative or baseline values); Test type: Superiority — We computed (post-hoc) the observed power of the performed tests (ANOVA for repeated measures). We confirmed that the specific sample size, as calculated using the Do-it-Yourself (DiY) quantitative research sample size calculator (available online at: https://blog.exmr.net/ sample-size-calculator) by considering a confidence level of 95% and a 10% margin of error, yielded adequate statistical power (> 80%) for each of the examined variables; p = 0.75, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 2: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.09, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 3: Comparison: Sham Bi-PAP vs Bi-PAP; 48 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.008, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 4: Comparison: Sham Bi-PAP vs Bi-PAP; 72 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.013, ANOVA — The a priori threshold for statistical significance was set at <0.05

3. Primary Outcome: Peak Expiratory Flow Rate (PEFR) Difference
Description: difference in PEFR value measured by spirometry pre- and post-operatively
Time Frame: 24 h before surgery and at 24, 48 and 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: Litres/minute
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
Litres/minute
  24h before surgery | 376.9 (71.7) | 325.3 (75.2)
  24h post-op | 146.9 (61.4) | 137.4 (30.5)
  48h post-op | 166.0 (68.1) | 195.7 (46.0)
  72h post-op | 190.1 (64.2) | 247.5 (60.5)
Statistical Analysis 1: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h before surgery (pre-operative or baseline values); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.05, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 2: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.55, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 3: Comparison: Sham Bi-PAP vs Bi-PAP; 48h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.13, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 4: Comparison: Sham Bi-PAP vs Bi-PAP; 72 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.011, ANOVA — The a priori threshold for statistical significance was set at <0.05

4. Primary Outcome: SpO2 Difference
Description: difference in SpO2 value measured by spirometry pre- and post-operatively
Time Frame: 24 h before surgery and at 24, 48 and 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
percentage of SpO2
  24h before surgery | 96.9 (0.7) | 96.9 (1.1)
  24h post-op | 91.6 (3.5) | 92.6 (3.2)
  48h post-op | 92.4 (3.5) | 95.2 (1.9)
  72h post-op | 92.5 (3.7) | 96.8 (1.0)
Statistical Analysis 1: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h before surgery (pre-operative or baseline values); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.83, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 2: Comparison: Sham Bi-PAP vs Bi-PAP; 24 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.37, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 3: Comparison: Sham Bi-PAP vs Bi-PAP; 48 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0035, ANOVA — The a priori threshold for statistical significance was set at <0.05
Statistical Analysis 4: Comparison: Sham Bi-PAP vs Bi-PAP; 72 h post-operatively; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.000015, ANOVA — The a priori threshold for statistical significance was set at <0.05

5. Primary Outcome: Number of Participants With Hypoxemia
Description: occurrence of hypoxemia, considered as SpO2<90%, post-operatively
Time Frame: At 24, 48 and 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
Participants
  24h post-op | 5 | 0
  48h post-op | 0 | 0
  72h post-op | 0 | 0

6. Primary Outcome: Number of Participants With Atelectasis
Description: occurrence of atelectasis as defined by chest X-ray (CXR) post-operatively with CXR before surgery as baseline
Time Frame: At 24, 48 and 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
Participants
  24h post-op | 3 | 0
  48h list-op | 3 | 0
  72h post-op | 3 | 0

7. Secondary Outcome: Post-operative Pain
Description: Intensity of pain was assessed post-operatively by Numerical Rating Scale (NRS) (0-10, 0=no pain, 10=worst pain imaginable)
Time Frame: right before spirometry, at 24, 48 and 72 h post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
score on a scale
  24h post-op | 6.5 (1.9) | 6.5 (1.3)
  48h post-op | 4.5 (1.5) | 5.3 (1.9)
  72h post-op | 3.3 (1.2) | 3.5 (1.4)

8. Secondary Outcome: Days of Hospitalization
Description: duration of hospitalization, calculated by discharge date minus admission date
Time Frame: From day of admission to day of discharge from the hospital
Population: Overall number of patients analyzed in each group is the sum of participants who underwent gastroplasty and those who underwent open gastric bypass (11+3=14 for the Sham Bi-PAP group and 15+6=21 for the Bi-PAP group).
Measure: Mean (Full Range); unit: days
Arm/Group | Sham Bi-PAP | Bi-PAP
Number analyzed (Participants) | 14 | 21
days
  Type of OBS: gastroplasty: number analyzed (Participants) | 11 | 15
  Type of OBS: gastroplasty | 6 [5 to 7] | 6 [5 to 7]
  Type of OBS: open gastric bypass: number analyzed (Participants) | 3 | 6
  Type of OBS: open gastric bypass | 10 [9 to 11] | 10 [9 to 11]

ADVERSE EVENTS:
Time Frame: Up to 1 year after study completion.
Arm/Group | Sham Bi-PAP | Bi-PAP
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 0/14 | 0/21

LIMITATIONS AND CAVEATS:
The small sample size in both groups, although calculated to provide adequate statistical power; low tolerance of the Bi-PAP device, which led to the exclusion of some subjects from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes